CLINICAL TRIAL: NCT05824689
Title: Exploratory Study of Fluoroquinolone Resistance for Patients Undergoing Autologous Hematopoietic Stem Cell (HSC) Transplantation in the Treatment of Multiple Myeloma
Brief Title: Fluoroquinolone Resistance Prevalence Study
Acronym: FRE
Status: Terminated | Type: Observational
Why Stopped: Discontinued Recruitment
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1263
Record Dates: First submitted 2023-03-24; First posted 2023-04-21 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
Keywords: Myeloma, Plasma-Cell; Fluoroquinolone resistance; Autologous Hematopoietic Stem Cell Transplantation; Antibiotic Prophylaxis; Gut Microbiome; Febrile neutropenia
MeSH Terms: conditions — Multiple Myeloma; Febrile Neutropenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an exploratory study to determine the prevalence of fluoroquinolone resistance in patients receiving dose-intense melphalan with autologous peripheral blood stem cell (PBSC) transplantation in the treatment of multiple myeloma (MM).

These data may be used in subsequent studies exploring the use of prophylaxis in this patient population.

DETAILED DESCRIPTION:
The goal of this observational study is to determine the prevalence of fluoroquinolone resistance in patients receiving dose-intense melphalan with autologous peripheral blood stem cell (PBSC) transplantation in the treatment of multiple myeloma (MM).

The main question[s] it aims to answer are:

* What is the prevalence of fluoroquinolone-resistant Enterobacterales (FRE) in patients undergoing autologous PBSC transplantation with dose-intense melphalan?
* Does the risk of febrile neutropenia differ in FRE carriers compared to non-carriers?

Participants will be tested for the presence of FRE before receiving fluoroquinolone prophylaxis at multiple points during the transplant course, including before chemotherapy mobilization (if used) using fluoroquinolone prophylaxis, at initial transplant hospitalization, at time of hospital discharge, and at or after day 84 after transplantation (day 0 is defined as day of HSC (hematopoietic stem cell) infusion).

FRE colonization will not be a determining factor in the use of fluoroquinolone prophylaxis during the treatment course.

This study will be open at two transplant units: Hackensack University Medical Center (HUMC) and MedStar Georgetown University Hospital (MGUH). Estimated number of subjects to be enrolled;

* HUMC: 124
* MGUH: 20

Anticipated enrollment period: 12-months with monitoring of subjects for 84 days (twelve weeks) after transplantation. Data will be analyzed over a three-month period (total study period of 18 months).

ELIGIBILITY:
Inclusion Criteria:

* Subjects >18 yrs of age.
* Diagnosis of multiple myeloma undergoing (first or subsequent) autologous PBSC transplantation.
* Transplant conditioning with melphalan 200 mg/m2.
* PBSC cell dose of >2x10e6 CD34+ cells/kg.
* Able to receive fluoroquinolone prophylaxis.
* Subjects must give consent for enrollment into this study.

Exclusion Criteria:

* Unwillingness to provide informed consent.
* Enrollment into a treatment protocol prescribing antibiotic prophylaxis.
* A diagnosis other than multiple myeloma.
* Receiving a conditioning regimen other than melphalan 200 mg/m2.
* Known light-chain amyloid deposition in any organ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects eligible for this study will meet the defined eligibility criteria to undergo autologous transplantation established at the transplant centers as per standard of care (SOC). All adult patients with a diagnosis of multiple myeloma undergoing autologous transplantation after dose-intense melphalan conditioning are candidates for enrollment into this study. These subjects will be approached for enrollment into this study by the transplant attending physician caring for the patient.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of FRE | Duration between Apheresis Consultation and Day +100
  Prevalence of FRE in patients undergoing autologous PBSC transplantation with dose-intense melphalan

SECONDARY OUTCOMES:
Occurrence/Risk of Febrile Neutropenia (FN) | Within 28 days of the transplantation
  Occurrence of neutropenic fever during the first 28 days (4 weeks) after autologous PBSC transplantation in the treatment of multiple myeloma.
Occurrence/Risk of Blood Stream infection (BSI) | Within 28 days of the transplantation
  The occurrence of Gram-negative BSI among the FRE carriers and FRE non-carriers
Comparison of severity of GI toxicity between FRE carriers and FRE non-carriers | Duration between Apheresis Consultation and Day +100
  Comparison of severity of GI toxicity between FRE carriers and FRE non-carriers per the grade of GI toxicity
Comparison of Length of Stay (LOS) between FRE carriers and FRE non-carriers | Duration between Day of hospital admission and Day of hospital discharge (estimated duration between 11 - 15 days)
  Comparison of Length of Stay (LOS) between FRE carriers and FRE non-carriers by estimating time to discharge
Comparison of Engraftment Kinetics between FRE carriers and FRE non-carriers | Duration between Apheresis Consultation and Day +100
  Comparison of Engraftment Kinetics (absolute neutrophil count (ANC), absolute lymphocyte count (ALC), platelet) between FRE carriers and FRE non-carriers

OTHER OUTCOMES:
Comparison of effect of FRE colonization and fluoroquinolone prophylaxis on the microbiome between FRE carriers and FRE non-carriers | Duration between Apheresis Consultation and Day +100
  Comparison of effect of FRE colonization and fluoroquinolone prophylaxis on the microbiome between FRE carriers and FRE non-carriers

CONTACTS AND LOCATIONS:
Overall Officials: Christina Cho, MD, Principal Investigator — Hackensack Meridian Health
Locations (2):
- United States (2):
  - Lombardi Comprehensive Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - John Theurer Cancer Center, Hackensack Meridian Health, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gafter-Gvili A, Fraser A, Paul M, Vidal L, Lawrie TA, van de Wetering MD, Kremer LC, Leibovici L. Antibiotic prophylaxis for bacterial infections in afebrile neutropenic patients following chemotherapy. Cochrane Database Syst Rev. 2012 Jan 18;1(1):CD004386. doi: 10.1002/14651858.CD004386.pub3. PMID 22258955
- [Background] Satlin MJ, Chen L, Douglass C, Hovan M, Davidson E, Soave R, La Spina M, Gomez-Arteaga A, van Besien K, Mayer S, Phillips A, Hsu JM, Malherbe R, Small CB, Jenkins SG, Westblade LF, Kreiswirth BN, Walsh TJ. Colonization With Fluoroquinolone-Resistant Enterobacterales Decreases the Effectiveness of Fluoroquinolone Prophylaxis in Hematopoietic Cell Transplant Recipients. Clin Infect Dis. 2021 Oct 5;73(7):1257-1265. doi: 10.1093/cid/ciab404. PMID 33956965
- [Background] Centers for Disease Control and Prevention; Infectious Diseases Society of America; American Society of Blood and Marrow Transplantation. Guidelines for preventing opportunistic infections among hematopoietic stem cell transplant recipients. Biol Blood Marrow Transplant. 2000;6(6a):7-83. doi: 10.1016/s1083-8791(00)70002-4. PMID 11185897
- [Background] Sorrig R, Klausen TW, Salomo M, Vangsted A, Gimsing P. Risk factors for infections in newly diagnosed Multiple Myeloma patients: A Danish retrospective nationwide cohort study. Eur J Haematol. 2019 Feb;102(2):182-190. doi: 10.1111/ejh.13190. Epub 2018 Nov 28. PMID 30485563
- [Background] Satlin MJ, Vardhana S, Soave R, Shore TB, Mark TM, Jacobs SE, Walsh TJ, Gergis U. Impact of Prophylactic Levofloxacin on Rates of Bloodstream Infection and Fever in Neutropenic Patients with Multiple Myeloma Undergoing Autologous Hematopoietic Stem Cell Transplantation. Biol Blood Marrow Transplant. 2015 Oct;21(10):1808-14. doi: 10.1016/j.bbmt.2015.06.017. Epub 2015 Jul 3. PMID 26150022
- [Background] Savage DG, Lindenbaum J, Garrett TJ. Biphasic pattern of bacterial infection in multiple myeloma. Ann Intern Med. 1982 Jan;96(1):47-50. doi: 10.7326/0003-4819-96-1-47. PMID 6976144
- [Background] Drayson MT, Bowcock S, Planche T, Iqbal G, Pratt G, Yong K, Wood J, Raynes K, Higgins H, Dawkins B, Meads D, Hulme CT, Monahan I, Karunanithi K, Dignum H, Belsham E, Neilson J, Harrison B, Lokare A, Campbell G, Hamblin M, Hawkey P, Whittaker AC, Low E, Dunn JA; TEAMM Trial Management Group and Trial Investigators. Levofloxacin prophylaxis in patients with newly diagnosed myeloma (TEAMM): a multicentre, double-blind, placebo-controlled, randomised, phase 3 trial. Lancet Oncol. 2019 Dec;20(12):1760-1772. doi: 10.1016/S1470-2045(19)30506-6. Epub 2019 Oct 23. PMID 31668592
- [Background] Sorrig R, Klausen TW, Salomo M, Vangsted A, Gimsing P. Risk factors for blood stream infections in multiple myeloma: A population-based study of 1154 patients in Denmark. Eur J Haematol. 2018 Jul;101(1):21-27. doi: 10.1111/ejh.13066. Epub 2018 May 4. PMID 29569379
- [Background] Jernigan JA, Hatfield KM, Wolford H, Nelson RE, Olubajo B, Reddy SC, McCarthy N, Paul P, McDonald LC, Kallen A, Fiore A, Craig M, Baggs J. Multidrug-Resistant Bacterial Infections in U.S. Hospitalized Patients, 2012-2017. N Engl J Med. 2020 Apr 2;382(14):1309-1319. doi: 10.1056/NEJMoa1914433. PMID 32242356
- [Background] Satlin MJ, Walsh TJ. Multidrug-resistant Enterobacteriaceae, Pseudomonas aeruginosa, and vancomycin-resistant Enterococcus: Three major threats to hematopoietic stem cell transplant recipients. Transpl Infect Dis. 2017 Dec;19(6):10.1111/tid.12762. doi: 10.1111/tid.12762. Epub 2017 Oct 25. PMID 28815897
- [Background] Spitzer TR. Engraftment syndrome following hematopoietic stem cell transplantation. Bone Marrow Transplant. 2001 May;27(9):893-8. doi: 10.1038/sj.bmt.1703015. PMID 11436099
- [Background] Maiolino A, Biasoli I, Lima J, Portugal AC, Pulcheri W, Nucci M. Engraftment syndrome following autologous hematopoietic stem cell transplantation: definition of diagnostic criteria. Bone Marrow Transplant. 2003 Mar;31(5):393-7. doi: 10.1038/sj.bmt.1703855. PMID 12634731
- [Background] Spitzer TR. Engraftment syndrome: double-edged sword of hematopoietic cell transplants. Bone Marrow Transplant. 2015 Apr;50(4):469-75. doi: 10.1038/bmt.2014.296. Epub 2015 Jan 12. PMID 25581406
- [Background] Gutierrez-Garcia G, Rovira M, Magnano L, Rosinol L, Bataller A, Suarez-Lledo M, Cibeira MT, de Larrea CF, Garrote M, Jorge S, Moreno A, Rodriguez-Lobato LG, Carreras E, Diaz-Ricart M, Palomo M, Martinez C, Urbano-Ispizua A, Blade J, Fernandez-Aviles F. Innovative strategies minimize engraftment syndrome in multiple myeloma patients with novel induction therapy following autologous hematopoietic stem cell transplantation. Bone Marrow Transplant. 2018 Dec;53(12):1541-1547. doi: 10.1038/s41409-018-0189-2. Epub 2018 Apr 29. PMID 29706650
- [Background] Chen J, Pan J, Zhan T, Tuazon S, Saini N, O'Hara W, Filicko-O'Hara J, Klumpp T, Kasner M, Carabasi M, Porcu P, Wagner JL. Autologous Stem Cell Transplantation for Multiple Myeloma: Growth Factor Matters. Biol Blood Marrow Transplant. 2019 Sep;25(9):e293-e297. doi: 10.1016/j.bbmt.2019.05.035. Epub 2019 Jun 4. PMID 31173899
- [Background] Ravoet C, Feremans W, Husson B, Majois F, Kentos A, Lambermont M, Wallef G, Capel P, Beauduin M, Delannoy A. Clinical evidence for an engraftment syndrome associated with early and steep neutrophil recovery after autologous blood stem cell transplantation. Bone Marrow Transplant. 1996 Nov;18(5):943-7. PMID 8932849
- [Background] Drobyski WR, Hari P, Keever-Taylor C, Komorowski R, Grossman W. Severe autologous GVHD after hematopoietic progenitor cell transplantation for multiple myeloma. Bone Marrow Transplant. 2009 Jan;43(2):169-77. doi: 10.1038/bmt.2008.295. Epub 2008 Sep 1. PMID 18762759
- [Background] Cornell RF, Hari P, Drobyski WR. Engraftment Syndrome after Autologous Stem Cell Transplantation: An Update Unifying the Definition and Management Approach. Biol Blood Marrow Transplant. 2015 Dec;21(12):2061-2068. doi: 10.1016/j.bbmt.2015.08.030. Epub 2015 Aug 29. PMID 26327628
- [Background] Rodriguez-Lobato LG, Martinez-Roca A, Castano-Diez S, Palomino-Mosquera A, Gutierrez-Garcia G, Pedraza A, Suarez-Lledo M, Rovira M, Martinez C, Fernandez de Larrea C, Cibeira MT, Rosinol L, Lozano E, Marin P, Cid J, Lozano M, Moreno-Castano AB, Palomo M, Diaz-Ricart M, Gallego C, Hernando A, Segura S, Carreras E, Urbano-Ispizua A, Blade J, Fernandez-Aviles F. The avoidance of G-CSF and the addition of prophylactic corticosteroids after autologous stem cell transplantation for multiple myeloma patients appeal for the at-home setting to reduce readmission for neutropenic fever. PLoS One. 2020 Nov 4;15(11):e0241778. doi: 10.1371/journal.pone.0241778. eCollection 2020. PMID 33147257
- [Background] Betticher C, Bacher U, Legros M, Zimmerli S, Banz Y, Mansouri Taleghani B, Pabst T. Prophylactic corticosteroid use prevents engraftment syndrome in patients after autologous stem cell transplantation. Hematol Oncol. 2021 Feb;39(1):97-104. doi: 10.1002/hon.2813. Epub 2020 Oct 3. PMID 32979278
- [Background] Shono Y, van den Brink MRM. Gut microbiota injury in allogeneic haematopoietic stem cell transplantation. Nat Rev Cancer. 2018 May;18(5):283-295. doi: 10.1038/nrc.2018.10. Epub 2018 Feb 16. PMID 29449660
- [Background] Van Lier YF, Van den Brink MRM, Hazenberg MD, Markey KA. The post-hematopoietic cell transplantation microbiome: relationships with transplant outcome and potential therapeutic targets. Haematologica. 2021 Aug 1;106(8):2042-2053. doi: 10.3324/haematol.2020.270835. PMID 33882637
- [Background] Peled JU, Devlin SM, Staffas A, Lumish M, Khanin R, Littmann ER, Ling L, Kosuri S, Maloy M, Slingerland JB, Ahr KF, Porosnicu Rodriguez KA, Shono Y, Slingerland AE, Docampo MD, Sung AD, Weber D, Alousi AM, Gyurkocza B, Ponce DM, Barker JN, Perales MA, Giralt SA, Taur Y, Pamer EG, Jenq RR, van den Brink MRM. Intestinal Microbiota and Relapse After Hematopoietic-Cell Transplantation. J Clin Oncol. 2017 May 20;35(15):1650-1659. doi: 10.1200/JCO.2016.70.3348. Epub 2017 Mar 15. PMID 28296584
- [Background] Samet A, Sledzinska A, Krawczyk B, Hellmann A, Nowicki S, Kur J, Nowicki B. Leukemia and risk of recurrent Escherichia coli bacteremia: genotyping implicates E. coli translocation from the colon to the bloodstream. Eur J Clin Microbiol Infect Dis. 2013 Nov;32(11):1393-400. doi: 10.1007/s10096-013-1886-9. Epub 2013 May 7. PMID 23649557
- [Background] Innes AJ, Mullish BH, Ghani R, Szydlo RM, Apperley JF, Olavarria E, Palanicawandar R, Kanfer EJ, Milojkovic D, McDonald JAK, Brannigan ET, Thursz MR, Williams HRT, Davies FJ, Marchesi JR, Pavlu J. Fecal Microbiota Transplant Mitigates Adverse Outcomes Seen in Patients Colonized With Multidrug-Resistant Organisms Undergoing Allogeneic Hematopoietic Cell Transplantation. Front Cell Infect Microbiol. 2021 Aug 27;11:684659. doi: 10.3389/fcimb.2021.684659. eCollection 2021. PMID 34513724
- [Background] Liao C, Taylor BP, Ceccarani C, Fontana E, Amoretti LA, Wright RJ, Gomes ALC, Peled JU, Taur Y, Perales MA, van den Brink MRM, Littmann E, Pamer EG, Schluter J, Xavier JB. Compilation of longitudinal microbiota data and hospitalome from hematopoietic cell transplantation patients. Sci Data. 2021 Mar 2;8(1):71. doi: 10.1038/s41597-021-00860-8. PMID 33654104
- [Background] El Jurdi N, Filali-Mouhim A, Salem I, Retuerto M, Dambrosio NM, Baer L, Lazarus HM, Caimi P, Cooper B, Tomlinson B, Metheny L, Malek E, Otegbeye F, Sekaly RP, Ghannoum M, de Lima M. Gastrointestinal Microbiome and Mycobiome Changes during Autologous Transplantation for Multiple Myeloma: Results of a Prospective Pilot Study. Biol Blood Marrow Transplant. 2019 Aug;25(8):1511-1519. doi: 10.1016/j.bbmt.2019.04.007. Epub 2019 Apr 5. PMID 30959164
- [Background] Khan N, Lindner S, Gomes ALC, Devlin SM, Shah GL, Sung AD, Sauter CS, Landau HJ, Dahi PB, Perales MA, Chung DJ, Lesokhin AM, Dai A, Clurman A, Slingerland JB, Slingerland AE, Brereton DG, Giardina PA, Maloy M, Armijo GK, Rondon-Clavo C, Fontana E, Bohannon L, Ramalingam S, Bush AT, Lew MV, Messina JA, Littmann E, Taur Y, Jenq RR, Chao NJ, Giralt S, Markey KA, Pamer EG, van den Brink MRM, Peled JU. Fecal microbiota diversity disruption and clinical outcomes after auto-HCT: a multicenter observational study. Blood. 2021 Mar 18;137(11):1527-1537. doi: 10.1182/blood.2020006923. PMID 33512409
- See also: Prevention and Treatment of Cancer-Related Infections, Version: 2.2020 — https://www.nccn.org